CLINICAL TRIAL: NCT06829888
Title: Percutaneous Tumor Ablation Versus Partial Nephrectomy for Small Renal Mass: the Impact of Histologic Variant and Tumor Size
Brief Title: Percutaneous Tumor Ablation Vs Partial Nephrectomy for Small Renal Mass: the Impact of Histologic Variant and Tumor Size
Acronym: CRYO-BO-2021
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: CRYO-BO-2021
Record Dates: First submitted 2025-01-10; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2024-12

CONDITIONS: Renal Cell Cancer
Keywords: Kidney neoplasms; Nephrectomy; Radiofrequency ablation; Cryosurgery; Recurrence
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- localized (cN0 M0) renal mass (cT1) treated with partial nephrectomy: patients with clinically localized (cN0 M0) renal mass (cT1) treated with partial nephrectomy
- localized (cN0 M0) renal mass (cT1) treated with percutaneus RFA: patients with clinically localized (cN0 M0) renal mass (cT1) treated with percutaneus RFA
- localized (cN0 M0) renal mass (cT1) treated with percutaneous cryo: patients with clinically localized (cN0 M0) renal mass (cT1) treated with percutaneous cryo

SUMMARY:
The aim, of this study is to investigate recurrence rates in patients with T1 renal cell carcinoma (RCC) undergone partial nephrectomy (PN), radiofrequency ablation (RFA) or cryoablation (Cryo).

DETAILED DESCRIPTION:
The aim of our study was to compare oncologic outcomes in terms of recurrence and competing causes of mortality in patients undergone either PN, radiofrequency ablation (RFA) or cryoablation (Cryo) focusing on tumor volume and histologic variant. Retrospectively were evaluated data from 665 (81.4%), 68 (8.3%) and 83 (10.3%) patients who underwent PN, RFA and Cryo, respectively. Kaplan-Meier curves depict recurrence-free survival (RFS) rates in the overall population and after stratifying according to tumor's histology (namely, clear cell RCC and non-clear RCC) and size (namely <2 cm and 2-4 cm). Multivariable Cox regression model was used to identify predictors of recurrence. Cumulative-incidence plots evaluated disease recurrence and other causes of mortality (OCM).

ELIGIBILITY:
Inclusion Criteria:

* Radiologic diagnosis (CT chest-abdomen or MRI abdomen with contrast medium) of renal neoplasm
* Renal neoplasm of clinical stage T1a (≤4 cm) N0M0
* Age >18 years
* Informed consent
* Absence of other neoplasm

Exclusion Criteria:

* Patients refuse partial nephrectomy and/or percutaneous renal CA and are candidates for active surveillance
* Patients who are candidates for radical nephrectomy

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data from 955 consecutive patients Were retrospectively selected with clinically localized (cN0 M0) renal mass (cT1) treated with PN or percutaneous RFA or percutaneous Cryo between January 2007 and July 2019.
  During preoperative workout, each patient performed either with abdominal and chest contrast enhanced computed tomography or magnetic resonance imaging to stage the disease. Tumor's complexity was defined according to PADUA score.11 Overall, 139 (14.6%) patients were excluded due to incomplete clinical data (Charlson Comorbidity Index [CCI], PADUA Score, clinical size of the tumor and age were lacking in 105 [10.9%], 75 [7.8%], 2 [0.2%] and2 [0.2%] patients, respectively), resulting in a final population of 816 individuals treated with PN (N.=665), RFA (N.=68) or Cryo (N.=83).
Sampling Method: Non-Probability Sample
Enrollment: 955 (Actual)
Dates: Start 2007-01-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
1. Disease recurrence of PN vs. RFA vs. Cryo after stratifying according to histological type and tumor size. | between January 2007 and July 2019
  No significant differences were recorded concerning the tumor's histology between the three groups. Patient follow-up for ablation was recommended at 3 months with abdominal CEUS and at 6 and 12 months with abdominal and chest CT or MRI followed by yearly intervals. In case of PN, the scheduled follow up included abdominal US at 6 months and abdominal and chest CT or MRI at 12 months, followed by two-yearly intervals. Local recurrence following ablation was defined as new focal enhancement in the ablation bed or enlargement of the ablation defect on follow-up imaging. Local recurrence following PN was defined as a mass in the ipsilateral kidney. Occurrence of metastatic disease was defined as extrarenal disseminated disease, with or without pathologic confirmation. Patients treated with PN experience better RFS rates as compared to both ablative techniques.However, considering patients with non-ccRCC and those with renal mass < 2cm, both PN and Cryo are valid options.

SECONDARY OUTCOMES:
Secondary outcome was death due to cause other than RCC (OCM) | between January 2007 and July 2019
  RCC was considered as the cause of death when it was registered as the first cause on death certificate, otherwise OCM was considered as the cause of death.PN proved to achieve better oncologic and survival outcomes compared to RFA and Cryo, since 91.2% vs. 67.8% and 60.2% of cases would be free from recurrence and OCM, respectively.These findings are mainly due to higher proportion of aged patients with shorter life expectancy in RFA and Cryo group than PN.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Bianchi, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna